CLINICAL TRIAL: NCT00455104
Title: Canadian Fabry Disease Initiative National Registry: Outcomes of Rare Disease Therapeutics and Cardiovascular Risk Factor Modification
Brief Title: Canadian Fabry Disease Initiative (CFDI) National Registry
Acronym: CFDI-NR
Status: Recruiting | Type: Observational
Sponsor: Canadian Fabry Research Consortium (Network)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: CFDI 001 - NR
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; National Registry
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Biomarker samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- National Registry: To maintain an established national registry which will collect information related to the identification and monitoring of all persons with Fabry disease in Canada.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational, voluntary registry.

SUMMARY:
CFDI NATIONAL REGISTRY

Fabry disease is a rare, inherited, genetic condition due to a deficiency of an enzyme called alpha-galactosidase A. This enzyme deficiency causes the small blood vessels to accumulate a substance called glycolipid. Without sufficient levels of the enzyme, alpha-galactosidase A, persons with Fabry Disease develop severe neuropathic pain, kidney disease, heart disease, stroke and/or premature death; often before the age of 60.

Fabry Disease is estimated to affect approximately one out of every 40,000 males and up to twice as many females in Canada. We do not have the exact number of persons in Canada who have this disease. A common problem in studying rare conditions is the difficulty in identifying the majority of people suffering from such a disease. Gathering their health information in order to better understand the natural disease progression and its response to treatment is difficult.

Early ERT studies involving humans had small numbers of subjects and the studies were of short duration. The results of these clinical studies did lead to approval of the therapy in many countries around the world including Canada. To date though, evidence of the usefulness of ERT and its direct impact on the natural course of Fabry disease has been limited, while its cost continues to be very high. As a result of these issues, there will need to be continued and long-term collection of information related to the effectiveness of ERT and other treatments to better document its true clinical outcomes in Canadian people with Fabry disease.

The Canadian Fabry Disease Initiative National Registry (CFDI-NR) is an observational, voluntary registry designed to collect outcomes data on Fabry disease from people living in Canada.

DETAILED DESCRIPTION:
CFDI NATIONAL REGISTRY: Canada-Wide Patient Recruitment

There are over 600 people in Canada known to have Fabry Disease. For more details about Fabry Disease, please refer to the "Brief Summary."

The goals of this nation-wide study are as follows:

1. To maintain an established national registry which will collect information related to the identification and monitoring of all persons with Fabry disease in Canada;
2. To determine clinical outcomes of patients with Fabry disease including those on treatment;
3. To determine if urine and plasma Gb3 and globotriasylsphingosine (LysoGb3) and their analogues can be biomarkers for Fabry disease and can predict clinical outcomes.

Data will be collected at baseline and every 12 months, as follows:

* Medical History
* Physical examination
* Neurological exam
* Electrocardiogram (ECG) - an electrical tracing of one's heart rhythm
* Echocardiogram (ultrasound of the heart)
* Holter monitor
* Magnetic Resonance Imaging (MRI) or CT Scan of the head
* Lab tests (including alpha-galactosidase levels)
* Review of current medications
* 24-hour urine collection or a random spot urine test
* Biomarker samples

To date though, evidence of the usefulness of ERT and its direct impact on the natural course of Fabry disease has been limited, while its cost continues to be very high (approximately $300,000 CDN per year per patient). As a result of these issues, there will need to be continued and long-term collection of information related to the effectiveness of ERT and other treatments to better document its true clinical outcomes in Canadian people with Fabry disease.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 5 years and older, up to & including age 85 years; and
* Able to give informed consent; and
* A clinical diagnosis of Fabry disease; and
* Compliance with all the clinic visits, interviews and assessments during the study period; and
* A Canadian citizen or a landed immigrant

EXCLUSION CRITERIA:

* Inability to give informed consent; or
* Problem complying with all the clinic visits, interviews and assessments during the study period; or
* An estimated life expectancy of less than 12 months
* Under 5 years of age
* Non-disease causing mutation

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Fabry disease living in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2007-01 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
(1) To maintain an established national database for the identification and monitoring of all patients with Fabry disease in Canada. | 2019

SECONDARY OUTCOMES:
2) To identify the clinical outcomes of patients with Fabry disease including those on various treatments. | 2019
3) To determine if urine and Gb3 and lysoGb3 and their analogues can be biomarkers for Fabry disease and can predict clinical outcomes. | 2019

CONTACTS AND LOCATIONS:
Overall Officials: Michael L West, MD, Principal Investigator — Queen Elizabeth II Health Sciences Centre (Capital District Health Authority), Halifax, Nova Scotia, Canada
Locations (5):
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - Vancouver General Hospital Adult Metabolic Diseases Clinic, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Toronto Western Hospital, Toronto, Ontario
  - University of Montreal, Department of Medicine, Montreal, Quebec

REFERENCES:
- See also: Fabry Disease: recommendations for diagnosis, management, and enzyme replacement therapy in Canada Nov 2005 — http://www.garrod.ca